CLINICAL TRIAL: NCT03311139
Title: Treatment and Outcomes Among Patients With Atrial Fibrillation and Acute Coronary Syndrome in Sweden
Brief Title: Treatment and Outcomes of Atrial Fibrillation and Acute Coronary Syndrome in Sweden
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 19562
Record Dates: First submitted 2017-09-28; First posted 2017-10-17 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Acute Coronary Syndrome; Anticoagulation
MeSH Terms: conditions — Atrial Fibrillation; Acute Coronary Syndrome | interventions — Fibrinolytic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AF and ACS patients: No PCI: Patients with Atrial Fibrillation and Acute Coronary Syndrom who did not undergo a Percutaneous Coronary Intervention
  Interventions: Drug: Antithrombotic agents
- AF and ACS patients: PCI without stent: Patients with Atrial Fibrillation and Acute Coronary Syndrom who underwent PCI without stent implantation (NOMESCO code FNG00-96 except FNG05)
  Interventions: Drug: Antithrombotic agents
- AF and ACS patients: PCI with stent: Patients with Atrial Fibrillation and Acute Coronary Syndrom who underwent PCI with stent implantation (NOMESCO code FNG05)
  Interventions: Drug: Antithrombotic agents

INTERVENTIONS:
Drug: Antithrombotic agents — Antiplatelets and anticoagulants purchased 4 months before and within 7 days after the index date

SUMMARY:
Many people who suffer from irregular heartbeats (atrial fibrillation) which might cause stroke, need to take blood thinners to prevent it. However, people with atrial fibrillation are also at increased risk of acute myocardial infarction or unstable angina pectoris (another heart condition marked by a chest pain, comprising so-called acute coronary syndrome for which another type of treatment that prevents blood from clotting (antiplatelet treatment) is indicated. In particularly if such patients undergo percutaneous coronary intervention, a procedure aimed to open up diseased blood vessels and hence to treat acute coronary syndrome, this treatment is needed. If a patients takes several anti-clotting blood drugs, the risk of bleeding is high. The number of possible drug combinations and treatment durations is large. This study will help us to understand which anti-clotting drug combinations are prescribed in real life among patients with atrial fibrillation and acute coronary syndrome, how effective and safe they are for patients. The study will look into the data that are already available in several very large Swedish databases which contain information needed for the research.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ACS defined by a hospital discharge (ICD-10 code of I21 for myocardial infarction or I20.0 for unstable angina pectoris (with or without sub-codes) during the study period and a diagnosis of AF (ICD-10 code I48 with or without sub-codes) in the Patient Register before or on the same day as the patient was discharged for ACS.

Exclusion Criteria:

- No exclusions will be made as the registries capture the entire life-time of entire population of Sweden.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population-based national Swedish dataset covering entire population without selection
Sampling Method: Non-Probability Sample
Enrollment: 14226 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Composition of treatment regimens | Minimum 3 months and up to 5 years and 1 month
  combinations of a vitamin K antagonist, antiplatelet therapy, a P2Y12 inhibitor without or with rivaroxaban in patients: who did not undergo Percutaneous Coronary Intervention (PCI), who underwent PCI without stent implantation (NOMESCO code FNG00-96 except FNG05), who underwent PCI with stent implantation (NOMESCO code FNG05).
Frequency of treatment regimens | Minimum 3 months and up to 5 years and 1 month
  frequency of identified drug combinations of a vitamin K antagonist, antiplatelet therapy, a P2Y12 inhibitor without or with rivaroxaban in patients: who did not undergo Percutaneous Coronary Intervention (PCI), who underwent PCI without stent implantation (NOMESCO code FNG00-96 except FNG05), who underwent PCI with stent implantation (NOMESCO code FNG05).
Prescribed strength of the most common regimens | Minimum 3 months and up to 5 years and 1 month
  prescribed strength of identified drug combinations of a vitamin K antagonist, antiplatelet therapy, a P2Y12 inhibitor without or with rivaroxaban in patients: who did not undergo Percutaneous Coronary Intervention (PCI), who underwent PCI without stent implantation (NOMESCO code FNG00-96 except FNG05), who underwent PCI with stent implantation (NOMESCO code FNG05)
Prescribed treatment duration of the most common regimens | Minimum 3 months and up to 5 years and 1 month
  prescribed duration of identified drug combinations of a vitamin K antagonist, antiplatelet therapy, a P2Y12 inhibitor without or with rivaroxaban in patients: who did not undergo Percutaneous Coronary Intervention (PCI), who underwent PCI without stent implantation (NOMESCO code FNG00-96 except FNG05), who underwent PCI with stent implantation (NOMESCO code FNG05)
Hospitalization or death with a diagnosis of bleeding as safety outcome | Minimum 3 months and up to 5 years and 1 month
  Total observation time is from 1st December 2011 and will include patients up to 31st December 2016. The analysis will be done in patients:
  who did not undergo Percutaneous Coronary Intervention (PCI), who underwent PCI without stent implantation (NOMESCO code FNG00-96 except FNG05), who underwent PCI with stent implantation (NOMESCO code FNG05)
Hospitalization for recurrent Acute Coronary Syndrom (ACS) as effectiveness outcome | Minimum 3 months and up to 5 years and 1 month
  Total observation time is from 1st December 2011 and will include patients up to 31st December 2016. The analysis will be done in patients:
  who did not undergo Percutaneous Coronary Intervention (PCI), who underwent PCI without stent implantation (NOMESCO code FNG00-96 except FNG05), who underwent PCI with stent implantation (NOMESCO code FNG05)
Revascularization procedure ( percutaneous stenting procedure or coronary bypass grafting) as effectiveness outcome | Minimum 3 months and up to 5 years and 1 month
  Total observation time is from 1st December 2011 and will include patients up to 31st December 2016. The analysis will be done in patients:
  who did not undergo Percutaneous Coronary Intervention (PCI), who underwent PCI without stent implantation (NOMESCO code FNG00-96 except FNG05), who underwent PCI with stent implantation (NOMESCO code FNG05)
Ischaemic stroke or systemic embolism as effectiveness outcome | Minimum 3 months and up to 5 years and 1 month
  Total observation time is from 1st December 2011 and will include patients up to 31st December 2016. The analysis will be done in patients:
  who did not undergo Percutaneous Coronary Intervention (PCI), who underwent PCI without stent implantation (NOMESCO code FNG00-96 except FNG05), who underwent PCI with stent implantation (NOMESCO code FNG05)
Death from any cause as effectiveness outcome | Minimum 3 months and up to 5 years and 1 month
  Total observation time is from 1st December 2011 and will include patients up to 31st December 2016. The analysis will be done in patients:
  who did not undergo Percutaneous Coronary Intervention (PCI), who underwent PCI without stent implantation (NOMESCO code FNG00-96 except FNG05), who underwent PCI with stent implantation (NOMESCO code FNG05)

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Sweden